CLINICAL TRIAL: NCT06112756
Title: A Randomized, Parallel-group Treatment, Phase 2, Double-blind Pilot Study to Investigate the Efficacy and Safety of Elinzanetant Compared With Placebo for Treatment of Sleep Disturbances Associated With Menopause.
Brief Title: A Study to Learn About How Elinzanetant Works and How Safe it is in Women Having Sleep Disturbances Associated With Menopause
Acronym: NIRVANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22423; 2023-504955-28-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Sleep Disturbances Associated With Menopause

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elinzanetant arm (Experimental): Participants will take Elinzanetant
  Interventions: Drug: Elinzanetant
- Placebo arm (Placebo Comparator): Participants will take elinzanetant matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Elinzanetant — Oral
  Arms: Elinzanetant arm
Other: Placebo — Oral
  Arms: Placebo arm

SUMMARY:
Researchers are looking for a better way to treat women who have sleep disturbances associated with menopause.

Menopause is part of a natural aging process and happens when women's menstrual cycles, also called periods, stop. Sleep disturbances, for example, frequent waking up at night, are a common and bothersome symptom associated with menopause that affects women's quality of life.

The study treatment Elinzanetant (also called BAY 3427080) is under development to treat symptoms like hot flashes which are caused by hormonal changes associated with menopause. It may block the activity of a protein that has been found to contribute to sleep disturbances.

The main purpose of this study is to learn how does elinzanetant affect sleep disturbances associated with menopause as measured on a sleep test called polysomnography (PSG) as compared with placebo.

For this, the researchers will analyze

* change in the total number of minutes a participant wakes up at night after going to sleep after 4 weeks of treatment compared to before treatment
* change in the total number of minutes a participant wakes up at night after going to sleep after 12 weeks of treatment compared to before treatment
* change in the participant's total time asleep while in bed after 4 and 12 weeks of treatment compared to before treatment.

The study participants will be randomly (by chance) assigned to one of two treatment groups. Dependent on the group, they will take elinzanetant or placebo for 12 weeks.

Each participant will be in the study for approximately 22 weeks (plus potential washout period), including a screening phase of up to 6 weeks, 12 weeks of treatment, and a follow up phase of 4 weeks after the end of treatment. 5 visits to the study site are planned.

During the study, the doctors and their study team will:

* take blood and urine samples
* do physical examinations
* check vital signs
* do sleep tests
* use an electronic hand-held device to record sleep quality and hot flashes at home

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40 to 65 years, inclusive, at signing of informed consent.
* Being in the post-menopausal period, defined as: serum FSH levels >40 mIU/mL and a serum estradiol concentration of <30 pg/mL at screening, AND Hysterectomy performed at least 6 weeks prior to screening.
* The participant's self-reported sleep history includes ongoing sleep disturbances associated with menopause characterized by waking up at night and/or poor quality of sleep.
* WASO of 30 minutes or more (mean of 2 screening PSGs with neither of the 2 nights <20 min).

Exclusion Criteria:

* Medical history, or baseline PSG assessment, includes a diagnosis of a sleep disorder other than sleep disturbances associated with the menopause (e.g., sleep apnea, restless leg syndrome, circadian rhythm sleep disorder).
* Current or history (except complete remission for 5 years or more) of any malignancy (except basal and squamous cell skin tumors).
* Renal impairment greater than moderate (i.e. estimated glomerular filtration rate <30 mL/min/1.73 m^2) at screening

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (22):
  - Preferred Research Partners, Little Port Walter, Alaska
  - MomDoc Women's Health Research | Scottsdale, AZ, Scottsdale, Arizona
  - Diagnamics | Encinitas, CA, Encinitas, California
  - SDS Clinical Trials Inc, Santa Ana, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - Helix Biomedics LLC | Boynton Beach, FL, Boynton Beach, Florida
  - Sweet Hope Research Specialty, Inc. - Hialeah, Hialeah, Florida
  - PharmaDev Clinical Research Institute, LLC, Miami, Florida
  - Segal Trials - Women's Health & General Medicine Research Site, North Miami, Florida
  - Palm Beach Research center, West Palm Beach, Florida
  - Sleep Practitioners, LLC, Macon, Georgia
  - SleepCare Research Institute Inc, Stockbridge, Georgia
  - Brengle Family Medicine, Indianapolis, Indiana
  - Revive Research Institute, Inc. - Women's Health, Dearborn Heights, Michigan
  - Essential Women's Health Associates, Las Vegas, Nevada
  - Clinilabs Drug Development Corporation-Feasibility, Eatontown, New Jersey
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, LLC., Cincinnati, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - FutureSearch Trials of Neurology LP, Austin, Texas
  - Sleep Therapy and Research Center | Medical Center Drive Office, San Antonio, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
- EMCO Privatklinik, Bad Dürrnberg, Salzburg, Austria
- Belgium (4):
  - Anima Research Center, Alken
  - SGS CPU, Edegem
  - Pneumocare SRL, Erpent
  - Universitair Ziekenhuis Leuven | Gasthuisberg Campus - Sleep Centre, Leuven
- Národní ústav duševního zdraví, Klecany, Czechia
- Germany (5):
  - Siteworks - Zentrum für klinische Studien Hannover, Hanover, Lower Saxony
  - Klinische Forschung Dresden | Dresden, Germany, Dresden, Saxony
  - ADVANCED SLEEP RESEARCH BERLIN Berlin, Berlin
  - KLIN FORSCHUNG HAMBURG GMBH Hamburg, Hamburg
  - SOMNI BENE INSTITUT FUR MEDIZIMISCHE FORSCHUNG & SCHLAFMEDEZIN Schwerin, Schwerin
- Poland (2):
  - Osrodek Medycyny Snu Instytutu Psychiatrii i Neurologii, Warsaw
  - EMC Instytut Medyczny SA, Wroclaw
- Spain (5):
  - Hospital Universitario de La Ribera | Neurophysiology and Sleep Department, Alzira
  - Centro Medico Teknon | Unidad de Medicina del Sueno, Barcelona
  - Hospital Clinico San Carlos | Neurophysiology Department - Sleep Unit - Menopause Sleep Disturbance, Madrid
  - Hospital Universitario HM Puerta Del Sur | Departamento de Ensayos Clinicos - Sleep Unit - Menopause Sleep Disturbance, Móstoles
  - Hospital Universitario de Araba | Santiago Campus - Unidad Sueno, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22423
- See also: US sites only: Click here for contact — https://www.probando.io/#/study-listing?CountryCode=us&SearchTerm=nirvana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 study centers, of which 30 centers had randomized participants in Europe and the US. In the US, separate sleep laboratories were used by 9 sites that did not have polysomnography (PSG) capability.
Pre-assignment Details: Out of the 338 screened participants, 110 were randomized and received treatment, and 103 participants completed the study. Among the 228 participants who did not proceed to randomization, screening failure was the primary reason (223 participants).
Groups:
- Elinzanetant: 120 mg (2x 60 mg soft gel capsules) of elinzanetant orally once daily for 12 weeks
- Placebo: 2 soft gel capsules orally once daily for 12 weeks
Period: Overall Study
Arm/Group | Elinzanetant | Placebo
Started | 55 | 55
Completed | 52 | 51
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Subject took an out of state job and had to early terminate | 1 | 0
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elinzanetant | Placebo | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (4.6) | 54.9 (4.7) | 54.8 (4.6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Only female participants enrolled
  Participants
    Female | 55 | 55 | 110
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 9 | 23
  White | 40 | 45 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Weight (kg) [Mean (Standard Deviation); unit: Kilograms] — Kilograms (Kg)
  Kilograms | 75.77 (12.45) | 74.41 (10.61) | 75.09 (11.53)
Height (cm) [Mean (Standard Deviation); unit: Centimeters] — Centimeters
  Centimeters | 164.64 (7.08) | 164.18 (7.01) | 164.41 (7.02)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: Kilogram per square meter] — Kilogram per square meter
  Kilogram per square meter | 27.97 (4.36) | 27.63 (3.75) | 27.80 (4.05)
Average weekly frequency of moderate to severe HF [Count of Participants; unit: Participants] — HF(s) Hot flash(es)
  Participants
    <35 moderate to severe HF per week | 13 | 11 | 24
    >=35 - <50 moderate to severe HF per week | 11 | 13 | 24
    >=50 moderate to severe HF per week | 31 | 31 | 62
Smoking [Count of Participants; unit: Participants]
  Never | 40 | 42 | 82
  Former | 5 | 10 | 15
  Current | 10 | 3 | 13
Alcohol consumption [Count of Participants; unit: Participants]
  Abstinent | 14 | 25 | 39
  Light | 41 | 30 | 71
Caffeine consumption (mg) per day [Mean (Standard Deviation); unit: Miligrams] | 142.07 (129.87) | 119.79 (99.53) | 131.43 (116.26)
Level of education [Count of Participants; unit: Participants]
  Missing | 1 | 0 | 1
  College or university education | 32 | 34 | 66
  Professional certification | 3 | 8 | 11
  Attending college | 5 | 3 | 8
  Other | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Wakefulness After Sleep Onset (WASO) at Week 4 as Measured by Polysomnography (PSG)
Description: WASO is defined as total time (min) spent awake from onset of persistent sleep to lights on.
  Persistent sleep is defined as 20 consecutive epochs (10 min) of non wakefulness. Smaller WASO values indicate shorter periods of wakefulness after sleep onset.
Time Frame: From baseline until week 4
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 47 | 47
Minutes | -23.50 (4.63) | -1.01 (4.68)

2. Secondary Outcome: Change From Baseline in WASO at Week 12 as Measured by PSG
Description: as for outcome 1
Time Frame: From baseline until week 12
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 46 | 43
Minutes | -16.48 (4.64) | -15.54 (4.76)

3. Secondary Outcome: Change From Baseline in Sleep Efficiency (SE) at Week 4 as Measured by PSG
Description: Sleep efficiency is defined as the percentage of time spent asleep while in bed. (Total sleep time / time in bed) x 100. Higher sleep efficiency values indicate more time spent asleep.
Time Frame: From baseline to Week 4
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 52 | 53
Percentage | 6.85 (8.07) | 1.13 (10.31)

4. Secondary Outcome: Change From Baseline in SE at Week 12 as Measured by PSG
Description: as for outcome 3
Time Frame: From baseline to week 12
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 52 | 51
Percentage | 5.15 (9.68) | 4.67 (8.10)

5. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) Total T-score at Week 4
Description: Participants' responses to the 8 items of the instrument are scored on a 1-5 numeric rating scale and will be aggregated to derive total raw scores ranging from 8-40 with higher scores indicating greater severity of sleep disturbance. These total raw scores will be converted into T-scores for comparison with population norms (United States general population). T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population.
Time Frame: From baseline until week 4
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 45 | 43
T-Score | -11.17 (8.04) | -6.59 (6.76)

6. Secondary Outcome: Change From Baseline inPatient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) Total T-score at Week 12
Description: as for outcome 5
Time Frame: From baseline until week 12
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 27 | 31
T-Score | -14.66 (9.36) | -6.65 (8.29)

7. Secondary Outcome: Change From Baseline in Insomnia Severity Index (ISI) Total Score at Week 4
Description: Insomnia Severity Index (ISI): The ISI is a 7-item tool that measures insomnia severity over the past two weeks (Bastien et al., 2001). It evaluates sleep onset, maintenance issues, early morning awakenings, satisfaction with sleep, noticeability of problems, distress caused, and daytime interference.
  Scoring: The ISI uses a 5-point Likert scale (0 to 4). Item scores are summed to yield a total score ranging from 0 to 28.
  Severity Categories:
  0-7: No clinically significant insomnia (better outcome) 8-14: Subthreshold insomnia (moderate outcome) 15-21: Clinical insomnia (moderate severity) (worse outcome) 22-28: Clinical insomnia (severe) (worse outcome) Interpretation: Higher total scores indicate worse insomnia severity, while lower scores indicate better sleep quality. The total score is the sum of individual item scores.
Time Frame: From baseline until week 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 48 | 50
Scores on a scale | -7.8 (6.0) | -4.7 (4.8)

8. Secondary Outcome: Change From Baseline in ISI Total Score at Week 12
Description: as for outcome 7
Time Frame: From baseline until week 12
Measure: Mean (Standard Deviation); unit: ISI total score
Arm/Group | Elinzanetant | Placebo
Number analyzed (Participants) | 42 | 47
ISI total score | -9.8 (6.4) | -6.9 (5.6)

ADVERSE EVENTS:
Time Frame: After the first study intervention up to 113 days until the last follow-up visit
Groups:
- BAY 3427080 / Elinzanetant: Soft gel capsule, two capsules of 60 mg
Arm/Group | BAY 3427080 / Elinzanetant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 2/55
Other Adverse Events (participants affected / at risk) | 24/55 | 25/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 3427080 / Elinzanetant (N=55) | Placebo (N=55)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 3427080 / Elinzanetant (N=55) | Placebo (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Thyroxine free increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (9) | 6 (7)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT06112756/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT06112756/SAP_001.pdf